CLINICAL TRIAL: NCT05683080
Title: The Impact of Achilles Tendon Rupture on the Structure and Function of the Achilles Tendon and Plantarflexors: a Longitudinal Cohort Study
Brief Title: Impact of Achilles Tendon Rupture on the Achilles Tendon and Calf Muscles
Acronym: ARCH
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0881
Record Dates: First submitted 2022-11-10; First posted 2023-01-12 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Achilles Tendon Rupture: Individuals who have experienced an Achilles tendon rupture and presented to the Achilles tendon rupture clinic.
  Interventions: Other: Routine Clinical Care

INTERVENTIONS:
Other: Routine Clinical Care — Participants completing the research study will receive routine clinical care

SUMMARY:
The aim of this study is to measure the recovery following Achilles tendon rupture. The investigators will use an ultrasound scan to look at the Achilles tendon, they will complete calf strength tests and use questionnaires to measure how individuals are managing in everyday life. The investigators will take these measurements when participants first arrive to the Achilles tendon rupture clinic, after 8 weeks, 10 weeks, 4 months, 6 months and 1 year.

DETAILED DESCRIPTION:
This study will measure the recovery of participants following Achilles tendon rupture. Measurements will be completed following Achilles tendon rupture, after 8 weeks, 10 weeks, 4 months, 6 months and 1 year. The measurements include an ultrasound tissue characterisation scan, isometric (static) strength test and heel raise test. In addition questionnaires will be completed by participants at each time point. Questionnaires include the Achilles Tendon Rupture Score, Hospital Anxiety and Depression Scale, EQ5D (a health related quality of life measure), International Physical Activity Questionnaire, Tampa Scale for Kinesiophobia and the Pain Catastrophising Scale.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* 16 years of age or above

Exclusion Criteria:

* Inability to provide informed consent due to cognitive impairment
* Inability to provide informed consent as unable to understand sufficient English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have experienced an Achilles Tendon Rupture and attended the Achilles Tendon Rupture Clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Ultrasound Tissue Characterisation | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  Imaging of the Achilles Tendon

SECONDARY OUTCOMES:
Change in Achilles Tendon Rupture Score | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  Scores are between 0-100 with a higher score indicating less severe limitations
Change in Hospital Anxiety and Depression Scale | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  The two domains (anxiety and depression) provide scores between 0-21 with a higher score indicating higher severity
Change in EuroQol- 5 Dimension -5 Level (EQ5D) | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  An index score is produced which is calculated using the UK index score reference. The thermometer score is between 0-100 with a higher score indicating better perceived health
Change in International Physical Activity Questionnaire | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or MET minutes representing the amount of energy expended carrying out physical activity. Higher METs indicate higher levels of physical activity
Change in Tampa Scale for Kinesiophobia | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia
Change in Pain Catastrophising Scale | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  A total score is calculated from 0-54 with a higher score indicating higher pain catastrophising
Change in Isometric plantarflexor strength testing | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  Isometric plantarflexor strength will be tested in plantargrade (neutral position) using the fysiometer.
Change in Heel Raise Test | Week 0, week8, week 10, 4 months, 6 months and 12 months
  The heel raise test will measure the amount of heel raises and the work completed by the participant in joules.
Change in 36-Item Short Form Survey (SF-36) | Week 0, week8, week 10, 4 months, 6 months and 12 months
  SF-36 measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). Higher scores indicate higher quality of life
Change in Activity Level | Week 0, week8, week 10, 4 months, 6 months and 12 months
  GENEactiv wrist based accelerometer measuring total steps, activity intensity 24 hours data capture for 7 days
Change in Sleep Duration | Week 0, week8, week 10, 4 months, 6 months and 12 months
  GENEactiv wrist based accelerometer measuring sleep duration for 7 days
Achilles Tendon Resting Angle | 12 month
  Measuring the resting angle of the achilles tendon

CONTACTS AND LOCATIONS:
Locations (1):
- University Hosptial of Leicester NHS Trust, Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No